CLINICAL TRIAL: NCT06636760
Title: Efficacy and Safety of Herbal Combination As Adjuvant Therapy for Mild and Moderate COVID-19 Patients
Brief Title: Efficacy and Immunomodulator Impact of Herbal Combination on COVID-19 Patients Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Anna Rozaliyani, M.Biomed, Sp.P(K), Department of Parasitology, Faculty of Medicine, Universitas Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-11-1403
Record Dates: First submitted 2024-09-26; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Herbal combination; Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Herbal Combination (Active Comparator)
  Interventions: Dietary Supplement: herbal compound

INTERVENTIONS:
Other: Placebo — The placebo contains the non-active carrier of herbal combination that has no pharmacological activity.
  Arms: Herbal combination; Placebo
Dietary Supplement: herbal compound — The herbal combination is made up of various medicinal plants and possesses immunomodulator properties. It comprises Phyllanthus niruri, Andrographis paniculata, and Glycyrrhiza glabra, along with Anacardium occidentale leaf and Zingiber officinale rhizome, all recognized for their immunomodulatory properties.
  Arms: Herbal Combination

SUMMARY:
This study aims to evaluate the efficacy and safety of Herbamuno+, a combination of several herbal ingredients, as an adjunct therapy for moderate COVID-19 patients at Wisma Atlet. The study involves 66 patients who were divided into two groups: one receiving Herbamuno+ and the other a placebo, both for 14 days. Researchers monitored clinical improvements, chest X-rays, and blood tests to assess inflammation and immune response. The goal is to determine whether Herbamuno+ can be safely and effectively added to standard COVID-19 treatment.

ELIGIBILITY:
Inclusion Criteria:

* The RCT included patients who met the following criteria: >18 years old, had recently tested positive for COVID-19 through RT-PCR within the past five days, and were categorized as moderate cases. The main clinical symptoms required for inclusion were acute fever (greater than 38 °C) and cough, or more than three of the following acute symptoms or signs: fever, cough, fatigue, headache, muscle pain, sore throat, nasal congestion, runny nose, shortness of breath, anorexia, nausea, vomiting, diarrhea, anosmia, or ageusia. The moderate case criteria are based on WHO criteria including the radiology imaging that indicating pneumonia (new infiltrates to consolidation) and clinical signs of pneumonia (fever, cough, shortness of breath, and respiratory frequency between 20 to 30 times per minute).

Exclusion Criteria:

* Patients were excluded if they had any of the following conditions: an oxygen saturation of less than 93%, participating in other clinical trials, pregnant or lactating, receiving other immunomodulatory drugs, had a history of allergies to the test product, or the history of tuberculosis, HIV/AIDS, psychosis, or autoimmune disorders. Subjects may also be dropped from the clinical trial if they withdraw, fail to comply with the protocol (including using less than 80% of the test product), disappear, or no longer meet the inclusion criteria. Adverse events, worsening conditions, or new diagnoses during the trial also warrant exclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Number of days required to improve clinical symptoms | 14 days
  This outcome measures how long it takes for a patient's symptoms to improve from the time of hospital admission based on anamnesis (patient history). Anamnesis includes information such as the duration and severity of the symptoms experienced by the patient. The improvement is tracked through daily assessments, comparing the patient's initial complaints upon admission to their status over time, noting any reduction in symptoms such as fever, cough, fatigue, or difficulty breathing. The goal is to quantify the days required to see a noticeable improvement in clinical symptoms.
Improvement of WHO ordinal scale | 14 days
  This outcome combines two critical assessments:
  WHO Ordinal Scale: This scale typically ranges from 0 (uninfected) to 8 (death), with each level corresponding to the patient's clinical status (e.g., mild disease, severe disease requiring oxygen support, or critical illness requiring mechanical ventilation). The improvement is measured by tracking the reduction in ordinal score over time, indicating a recovery or a shift toward a less severe category.
The EQ-5D-5L Quality of Life Measure | 14 days
  The EQ-5D-5L covers five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and has five response levels for each dimension, ranging from no problems to extreme problems. Improvement in this measure indicates better overall health and well-being. The EQ-5D-5L also includes a visual analog scale (VAS) where patients rate their overall health from 0 (worst possible health) to 100 (best possible health).
Number of days required for respiratory rate to return to normal | 14 days
  This outcome measures how long the patient's respiratory rate stabilizes and returns to normal levels. A normal respiratory rate in adults is typically 12 to 20 breaths per minute. This measure focuses on how many days it takes for the respiratory rate to reduce to or below 20 breaths per minute (indicating improvement from conditions such as tachypnea or labored breathing). Daily monitoring is required to track this change, as an elevated respiratory rate is a common symptom of respiratory distress, infection, or severe illness.

CONTACTS AND LOCATIONS:
Locations (1):
- The National Emergency Hospital for COVID-19, Wisma Atlet, Jakarta, DKI Jakarta, Indonesia